CLINICAL TRIAL: NCT01966068
Title: Informing Policy to Implement Pediatric Family Engagement in Meaningful Use Stage 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); American Academy of Pediatrics (Other); DARTNet Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-010285
Record Dates: First submitted 2013-10-11; First posted 2013-10-21 (Estimated); Results first posted 2016-08-30 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: Asthma; Pediatrics; Health Technology; Meaningful Use Stage-3; Web Portal
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MyAsthma Web Portal (Experimental): The portal, MyAsthma, will provide asthma education, collect patient-reported outcomes, evaluate medication use and side effects, and track parents' concerns and goals. Parents will log into the web portal each month (for a total of 3 portal visits in 6 months), and the information entered by parents will be shared through the electronic health record with the child's primary care provider.
  Interventions: Other: MyAsthma Web Portal

INTERVENTIONS:
Other: MyAsthma Web Portal — Parents will log on to the MyAsthma Web Portal up to three different times over a 6 month period. During each portal visit, parents will be asked to complete a survey which will include questions regarding their views on treatment preferences, goals, asthma control, and medications for their child with asthma.

SUMMARY:
This study will enroll parents/guardians of children who receive treatment at one of the pediatric primary care practice settings in the Pediatric Research in Office Settings (PROS) network or at the Children's Hospital of Philadelphia's Pediatric Research Consortium (PeRC) network.

The study will use an evidence-based conceptual model to study determinants of implementation success, implementation outcomes, and health care outcomes resulting from implementing an already functional, electronic health record (EHR)-linked asthma portal, MyAsthma. The study will measure the portal's feasibility and determine the impact on providing asthma education and fostering patient engagement as well as the ability to collect patient-reported outcomes for children, evaluate medication use and side effects and track parents' preferences and goals.

DETAILED DESCRIPTION:
This study uses a newly published, evidence-based conceptual model to study the determinants of implementation success, implementation outcomes, and health care outcomes resulting from implementing an asthma portal, MyAsthma, in the national, Agency for Health Care Research and Quality(AHRQ)-funded, Center for Pediatric Practice Research and Learning. Technically, the portal will be implemented with 2 innovative approaches that facilitate rapid cycle evaluation in multiple Electronic Health Records (EHRs). Although many patient portals are simple vehicles for transferring information about upcoming appointments, test results or laboratory findings, the asthma portal in this project extends this basic functionality to provide asthma education, collect patient-reported outcomes, evaluate medication use and side effects, and track parents' preferences and goals. Because asthma is an AHRQ priority condition which addresses three AHRQ priority criteria (children, low income, and special health care needs), our study will use this population to focus on stage 3 Meaningful Use (MU3) objectives. It is the hope that by conducting this study, translational knowledge will be gained to make recommendations for practice implementation and actionable policy statements.

ELIGIBILITY:
Inclusion Criteria For Parents/Guardians:

1. Parent/guardian of a child who:

   * Is between the ages of 6-12 years old
   * Has a diagnosis of asthma on his/her problem list at the time of recruitment
   * Has had an office visit with asthma as a diagnosis within the past 12 months
2. Must be able to speak and read English

Exclusion Criteria For Parents/Guardians:

1. Child has not had an office visit for asthma with in the last 12 months
2. Parent or guardian does not speak or read English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Pediatrick Research in Office Settings (PROS), Elk Grove Village, Illinois
  - Pediatric Research Consortium of the Children's Hospital of Philadelphia (PeRC), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fiks AG, DuRivage N, Mayne SL, Finch S, Ross ME, Giacomini K, Suh A, McCarn B, Brandt E, Karavite D, Staton EW, Shone LP, McGoldrick V, Noonan K, Miller D, Lehmann CU, Pace WD, Grundmeier RW. Adoption of a Portal for the Primary Care Management of Pediatric Asthma: A Mixed-Methods Implementation Study. J Med Internet Res. 2016 Jun 29;18(6):e172. doi: 10.2196/jmir.5610. PMID 27357835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2 practice-based research networks. To ensure low-income children were represented, practices were required to have at least 20% insured by Medicaid or the Children's Health Insurance Program. 9,133 families were invited to enroll.
Pre-assignment Details: 294 parents/guardians of 294 children consented to participate in the study. Of these, 237 logged onto the MyAsthma portal at least once.
Groups:
- MyAsthma Web Portal: The portal, MyAsthma, provided asthma education, collected patient-reported outcomes, evaluated medication use and side effects, and tracked parents' concerns and goals. Parents logged into the web portal each month, and the information entered by parents was shared through the electronic health record with the child's primary care provider.
Period: Overall Study
Arm/Group | MyAsthma Web Portal
Started | 294
Used the MyAsthma Portal at Least Once | 237
Use the MyAsthma Portal More Than Once | 156
Completed | 156
Not Completed | 138
Not completed — Withdrawal by Subject | 57
Not completed — Lost to Follow-up | 81

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included every family of children with asthma who logged onto the MyAsthma portal at least once.
Groups:
- MyAsthma Web Portal Sustained Use: Subject (parent/guardian) logged on to the MyAsthma Web Portal and completed surveys more than once
- MyAsthma Web Portal Adoption: Subject (parent/guardian) logged on to the MyAsthma Web Portal and completed surveys only once
- Total: Total of all reporting groups
Arm/Group | MyAsthma Web Portal Sustained Use | MyAsthma Web Portal Adoption | Total
Number analyzed (Participants) | 156 | 81 | 237
Age, Continuous [Mean (Standard Deviation); unit: years] — Parent's Age
  years | 38.1 (5.5) | 37.1 (6.5) | 37.6 (6.0)
Age, Customized [Number; unit: participants] — Child's Age
  participants
    6-9 Years | 115 | 60 | 175
    10-12 Years | 41 | 21 | 62
Sex: Female, Male [Count of Participants; unit: Participants] — Child's Gender
  Participants
    Female | 71 | 30 | 101
    Male | 85 | 51 | 136
Race/Ethnicity, Customized [Number; unit: participants] — Parent's Race
  participants
    White | 93 | 55 | 148
    Black/African American | 48 | 20 | 68
    Asian | 4 | 0 | 4
    Other | 11 | 6 | 17
Race/Ethnicity, Customized [Number; unit: participants] — Child's Race
  participants
    White | 89 | 55 | 144
    Black/African American | 54 | 21 | 75
    Asian | 4 | 0 | 4
    Other | 7 | 4 | 11
    Unkown | 2 | 1 | 3
Parent Education [Number; unit: participants]
  High School or Less | 17 | 17 | 34
  Some College/Associates | 46 | 35 | 81
  Bachelor's or Higher | 93 | 29 | 122
Parent Employment Status [Number; unit: participants]
  Working Outside the Home | 111 | 46 | 157
  Self-Employed | 5 | 8 | 13
  Working Without Pay | 25 | 18 | 43
  Unemployed | 15 | 9 | 24
Parent's Relation to Child [Number; unit: participants]
  Mother | 149 | 79 | 228
  Other | 7 | 2 | 9
Child's Asthma Severity [Number; unit: participants]
  Intermittent | 37 | 12 | 49
  Mild Persistent | 39 | 12 | 51
  Moderate/Severe Persistent | 17 | 2 | 19
  Unknown | 63 | 55 | 118
Medical Practice Setting [Number; unit: participants]
  Urban | 44 | 20 | 64
  Rural | 29 | 23 | 52
  Suburban | 83 | 38 | 121

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Number of Families Who Adopted MyAsthma Portal Use and Number of Families With Sustained Use
Description: Implementation success was measure by comparing the of the number of enrolled families (parent/guardian) who logged on to the MyAsthma Portal once (adoption) with the number of enrolled families (parent/guardian) who logged on more than once (sustained use). Parents/guardians were asked to log on and complete the same survey on the MyAsthma Portal 3 times during a 6 month period.
Time Frame: Up to 6 Months
Population: Analysis population included every subject (parent/guardian) who logged on to the MyAsthma Web Portal at least once.
Measure: Number; unit: participants
Groups:
- MyAsthma Portal Adoption: Subject (parent/guardian) logged on to the MyAsthma Web Portal and completed surveys only once.
Arm/Group | MyAsthma Web Portal Sustained Use | MyAsthma Portal Adoption
Number analyzed (Participants) | 237 | 237
participants | 156 | 81

ADVERSE EVENTS:
Time Frame: 6 Months
Groups:
- MyAsthma Web Portal: The portal, MyAsthma, will provide asthma education, collect patient-reported outcomes, evaluate medication use and side effects, and track parents' concerns and goals. Parents will log into the web portal each month, and the information entered by parents will be shared through the electronic health record with the child's primary care provider.
  MyAsthma Web Portal
Arm/Group | MyAsthma Web Portal
Serious Adverse Events (participants affected / at risk) | 0/237
Other Adverse Events (participants affected / at risk) | 0/237

LIMITATIONS AND CAVEATS:
Enrollment occurred in practices across 11 states, yet more than half of practices were within a single health system thus affecting generalizability. This study also includes a relatively short follow-up period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes